CLINICAL TRIAL: NCT06025201
Title: Characterization of Longitudinal EEG Biomarkers in Chronic Low Back Pain
Brief Title: Detection of EEG-Based Biomarkers of Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Edward Lannon, Pain Psychologist, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 71778; 1K23AR083171-01 (NIH)
Record Dates: First submitted 2023-08-24; First posted 2023-09-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain; Healthy

STUDY DESIGN:
Intervention Model Description: All participants will complete all interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All participants will complete all interventions
  Interventions: Behavioral: Resting State EEG; Behavioral: Picture Viewing EEG; Behavioral: Stop Signal EEG

INTERVENTIONS:
Behavioral: Resting State EEG — During this intervention, participants will be asked to not think about anything in particular while EEG is recorded. Resting state will be conducted with either the participants having their eyes open, or eyes closed.
Behavioral: Picture Viewing EEG — During this intervention, participants will view emotionally charged pictures for a short period of time. Afterwards, participants will be asked to rate their emotional reactions to the pictures. EEG will be recorded during this intervention.
Behavioral: Stop Signal EEG — During this intervention, participants will be asked to respond quickly to a visual stimulus with a button press. At times, participants will be asked to inhibit their responses. EEG will be recorded during this intervention.

SUMMARY:
Chronic low back pain (CLBP) is a pervasive disorder affecting up to one-fifth of adults globally and is the single greatest cause of disability worldwide. Despite the high prevalence and detrimental impact of CLBP, its treatments and mechanisms remain largely unclear. Biomarkers that predict symptom progression in CLBP support precision-based treatments and ultimately aid in reducing suffering. Longitudinal brain-based resting-state neuroimaging of patients with CLBP has revealed neural networks that predict pain chronification and its symptom progression. Although early findings suggest that measurements of brain networks can lead to the development of prognostic biomarkers, the predictive ability of these models is strongest for short-term follow-up. Measurements of different neural systems may provide additional benefits with better predictive power.

Emotional and cognitive dysfunction is common in CLBP, occurring at the behavioral and cerebral level, presenting a unique opportunity to detect prognostic brain-based biomarkers. Likewise, improvements in electroencephalogram (EEG) neuroimaging strategies have led to increased spatial resolution, enabling researchers to overcome the limitations of classically used neuroimaging modalities (e.g., magnetic resonance imaging [MRI] and functional MRI), such as high cost and limited accessibility. Using longitudinal EEG, this patient-oriented research project will provide a comprehensive neural picture of emotional, cognitive, and resting-state networks in patients with CLBP, which will aid in predicting symptom progression in CLBP. Through this award, the investigators will use modern EEG source analysis strategies to track biomarkers at baseline and 1- and 2-month follow-ups and their covariance with markers for pain and emotional and cognitive dysfunction. A 5-month follow up will also be used to only assess patient reported outcomes. In Aim 1, the investigators will identify and characterize differences in resting-state, emotional, and cognitive networks between patients with CLPB and age/sex-matched controls. In Aim 2, the investigators will identify within-subject changes across time and their relationship with clinical symptoms. In Aim 3, as an exploratory aim, the investigators will apply machine- and deep-learning strategies to detect a comprehensive signature of CLBP using EEG features from resting-state, emotional, and cognitive networks.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Chronic Low Back Pain

Exclusion Criteria:

* Current diagnosis of cancer
* Severe psychiatric conditions
* Pending personal litigation relating to an injury or receiving workers' compensation benefits
* Being a non-English speaker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity changes from baseline as assessed by the PROMIS current, 7 day maximal and 7 day average | Baseline, 1-month, 2-month and 5-month follow-ups
  Within subjects change in pain intensity from baseline to each follow up point. Pain intensity measures are 0-10 range with larger numbers indicating more pain
EEG resting state functional connectivity changes from baseline | Baseline, 1-month and 2-month follow-ups
  Within subjects change in resting state functional connectivity from baseline to each follow up point.
EEG late positive potential changes from baseline | Baseline, 1-month and 2-month follow-ups
  Within subjects change in late positive potential from baseline to each follow up point.
EEG error related negativity changes from baseline | Baseline, 1-month and 2-month follow-ups
  Within subjects change in error related negativity from baseline to each follow up point.

SECONDARY OUTCOMES:
Neuropsychological changes from baseline as assessed by the NIH toolbox | Baseline, 1-month and 2-month follow-ups
  Within subjects change in metrics of fluid and crystallized intelligence from baseline to each follow up point

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford's Systems and Neuroscience Pain Lab, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will support requests for data sharing in a timely manner. Prior to sharing data, the data will be redacted of all personal identifiers to prevent subject identification.